CLINICAL TRIAL: NCT02660242
Title: The Use of Mini-dose Glucagon to Prevent Exercise-induced Hypoglycemia in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Xeris Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: T1DX Mini-dose Exercise
Record Dates: First submitted 2016-01-06; First posted 2016-01-21 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; Type 1 Diabetes; Mini-dose Glucagon; Adults; Exercise; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): No basal insulin adjustment, no carbohydrate intake (until glucose drops <70 mg/dL).
- Basal insulin reduction (Active Comparator): Basal insulin reduction to 50% five minutes before the start of exercise.
  Interventions: Other: Basal Insulin Reduction
- Glucose Tabs (Active Comparator): Dextrose tabs orally (20 grams) five minutes before the start of exercise and at 30 minutes of exercise (total 40 grams).
  Interventions: Other: Glucose Tabs
- G-Pen Mini™ (glucagon injection) (Experimental): Glucagon (150 µg) five minutes before the start of exercise (SQ-abdomen).
  Interventions: Drug: G-Pen Mini™ (glucagon injection)

INTERVENTIONS:
Drug: G-Pen Mini™ (glucagon injection) — Glucagon (150 µg) 5 minutes before the start of exercise (SQ-abdomen).
  Other Names: mini-dose glucagon
  Arms: G-Pen Mini™ (glucagon injection)
Other: Glucose Tabs — Dextrose tabs orally (20 grams) 5 minutes before the start of exercise and at 30 minutes of exercise (total 40 grams).
  Other Names: over-the-counter oral glucose tablets
  Arms: Glucose Tabs
Other: Basal Insulin Reduction — Basal insulin reduction to 50% 5 minutes before the start of exercise.
  Arms: Basal insulin reduction

SUMMARY:
This project focuses on development of new strategy for the prevention of exercise-associated hypoglycemia using mini-dose glucagon.

DETAILED DESCRIPTION:
The primary objective of the protocol is to determine if the administration of mini-dose glucagon administered subcutaneously just before exercise produces better glucose stability than no adjustments for moderate intensity exercise in patients with Type 1 Diabetes (T1D). It will also be assessed whether mini-dose glucagon before exercise produces better glucose stability than basal insulin reductions or extra carbohydrate consumption.

This is a randomized, 4-way crossover trial. The trial will include 16 participants who complete the study.

Each participant will undergo four aerobic exercise sessions (in random order), with different strategies for glucose regulation:

* Control Trial: Fasted exercise, no basal insulin reduction
* Strategy 1: Fasted exercise, basal insulin reduction only (50% reduction in basal rate at 60 minutes before exercise, for the duration of the exercise)
* Strategy 2: Fasted exercise, no basal adjustment + pre-exercise glucose tabs (buccal route-40 grams in total )
* Strategy 3: Fasted exercise, no basal adjustment + pre-exercise mini-dose glucagon (sc)

In all 4 sessions, aerobic exercise will be performed in the fasted state (before a standardized meal) for 45 minuets at ~50-55% of the participant's per-determined aerobic capacity. The participant's pump will be blinded during the control trial, strategy 1, and strategy 3 and an injection of saline will be given during the control trial and strategy 1 so that participant is blinded to strategy.

The primary outcome for this study will be the glycemic response during exercise and early recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of presumed autoimmune type 1 diabetes, receiving daily insulin
2. Age 18-<65 years
3. Duration of T1D ≥ 2 years
4. Random C-peptide < 0.6 ng/ml
5. Using continuous subcutaneous insulin infusion (CSII; insulin pump) for at least 6 months, with no plans to discontinue pump use during the study
6. Exercises regularly, i.e. ≥30 minutes moderate or more vigorous aerobic activity X ≥3 times/week
7. Body mass index (BMI) <30 kg/m2
8. Females must meet one of the following criteria:

   * Of childbearing potential and not currently pregnant or lactating, and agrees to use an accepted contraceptive regimen as described in the study procedure manual throughout the entire duration of the study; or
   * Of non-childbearing potential, defined as a female who has had a hysterectomy or tubal ligation, is clinically considered infertile or is in a menopausal state (at least 1 year without menses)
9. In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
10. Willing to adhere to the protocol requirements for the duration of the study
11. Must be enrolled in the T1D Exchange clinic registry or willing to join the registry

Exclusion Criteria:

1. One or more severe hypoglycemic episodes in the past 12 months (as defined by an episode that required third party assistance for treatment)
2. Active diabetic retinopathy (proliferative diabetic retinopathy or vitreous hemorrhage in past 6 months) that could potentially be worsened by exercise protocol
3. Peripheral neuropathy with insensate feet
4. Cardiovascular autonomic neuropathy with inappropriate heart rate response to exercise
5. Use of non-insulin anti-diabetic medications
6. Use of beta-blockers
7. Use of agents that affect hepatic glucose production such as beta adrenergic agonists, xanthine derivatives
8. Use of Pramlintide
9. Currently following a very low calorie or other weight-loss diet
10. Participation in other studies involving administration of an investigational drug or device within 30 days or 5 half-lives, whichever is longer, before screening for the current study or planning to participate in another such study during participation in the current study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Riddell, PhD, Study Chair — York University; Michael Rickels, M.D., M.S., Study Chair — University of Pennsylvania; Howard Wolpert, M.D., Study Chair — Joslin Diabetes Center; Stephanie DuBose, M.P.H, Principal Investigator — Jaeb Center for Health Research
Locations (2):
- United States (2):
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Chu L, Hamilton J, Riddell MC. Clinical management of the physically active patient with type 1 diabetes. Phys Sportsmed. 2011 May;39(2):64-77. doi: 10.3810/psm.2011.05.1896. PMID 21673486
- [Background] West DJ, Morton RD, Bain SC, Stephens JW, Bracken RM. Blood glucose responses to reductions in pre-exercise rapid-acting insulin for 24 h after running in individuals with type 1 diabetes. J Sports Sci. 2010 May;28(7):781-8. doi: 10.1080/02640411003734093. PMID 20496226
- [Background] Brazeau AS, Rabasa-Lhoret R, Strychar I, Mircescu H. Barriers to physical activity among patients with type 1 diabetes. Diabetes Care. 2008 Nov;31(11):2108-9. doi: 10.2337/dc08-0720. Epub 2008 Aug 8. PMID 18689694
- [Background] Rabasa-Lhoret R, Bourque J, Ducros F, Chiasson JL. Guidelines for premeal insulin dose reduction for postprandial exercise of different intensities and durations in type 1 diabetic subjects treated intensively with a basal-bolus insulin regimen (ultralente-lispro). Diabetes Care. 2001 Apr;24(4):625-30. doi: 10.2337/diacare.24.4.625. PMID 11315820
- [Background] Campbell MD, Walker M, Trenell MI, Jakovljevic DG, Stevenson EJ, Bracken RM, Bain SC, West DJ. Large pre- and postexercise rapid-acting insulin reductions preserve glycemia and prevent early- but not late-onset hypoglycemia in patients with type 1 diabetes. Diabetes Care. 2013 Aug;36(8):2217-24. doi: 10.2337/dc12-2467. Epub 2013 Mar 20. PMID 23514728
- [Background] Stenerson M, Cameron F, Payne SR, Payne SL, Ly TT, Wilson DM, Buckingham BA. The impact of accelerometer use in exercise-associated hypoglycemia prevention in type 1 diabetes. J Diabetes Sci Technol. 2015 Jan;9(1):80-5. doi: 10.1177/1932296814551045. Epub 2014 Sep 17. PMID 25231116
- [Background] Tsalikian E, Mauras N, Beck RW, Tamborlane WV, Janz KF, Chase HP, Wysocki T, Weinzimer SA, Buckingham BA, Kollman C, Xing D, Ruedy KJ; Diabetes Research In Children Network Direcnet Study Group. Impact of exercise on overnight glycemic control in children with type 1 diabetes mellitus. J Pediatr. 2005 Oct;147(4):528-34. doi: 10.1016/j.jpeds.2005.04.065. PMID 16227041
- [Background] Tanenberg RJ, Newton CA, Drake AJ. Confirmation of hypoglycemia in the "dead-in-bed" syndrome, as captured by a retrospective continuous glucose monitoring system. Endocr Pract. 2010 Mar-Apr;16(2):244-8. doi: 10.4158/EP09260.CR. PMID 19833577
- [Background] Campbell MD, Walker M, Trenell MI, Luzio S, Dunseath G, Tuner D, Bracken RM, Bain SC, Russell M, Stevenson EJ, West DJ. Metabolic implications when employing heavy pre- and post-exercise rapid-acting insulin reductions to prevent hypoglycaemia in type 1 diabetes patients: a randomised clinical trial. PLoS One. 2014 May 23;9(5):e97143. doi: 10.1371/journal.pone.0097143. eCollection 2014. PMID 24858952
- [Background] Taplin CE, Cobry E, Messer L, McFann K, Chase HP, Fiallo-Scharer R. Preventing post-exercise nocturnal hypoglycemia in children with type 1 diabetes. J Pediatr. 2010 Nov;157(5):784-8.e1. doi: 10.1016/j.jpeds.2010.06.004. Epub 2010 Jul 21. PMID 20650471
- [Background] Riddell MC, Bar-Or O, Ayub BV, Calvert RE, Heigenhauser GJ. Glucose ingestion matched with total carbohydrate utilization attenuates hypoglycemia during exercise in adolescents with IDDM. Int J Sport Nutr. 1999 Mar;9(1):24-34. doi: 10.1123/ijsn.9.1.24. PMID 10036339
- [Background] Robertson K, Riddell MC, Guinhouya BC, Adolfsson P, Hanas R; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Exercise in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:203-23. doi: 10.1111/pedi.12176. No abstract available. PMID 25182315
- [Background] Camacho RC, Galassetti P, Davis SN, Wasserman DH. Glucoregulation during and after exercise in health and insulin-dependent diabetes. Exerc Sport Sci Rev. 2005 Jan;33(1):17-23. PMID 15640716
- [Background] Oskarsson PR, Lins PE, Wallberg Henriksson H, Adamson UC. Metabolic and hormonal responses to exercise in type 1 diabetic patients during continuous subcutaneous, as compared to continuous intraperitoneal, insulin infusion. Diabetes Metab. 1999 Dec;25(6):491-7. PMID 10633873
- [Background] Haymond MW, Schreiner B. Mini-dose glucagon rescue for hypoglycemia in children with type 1 diabetes. Diabetes Care. 2001 Apr;24(4):643-5. doi: 10.2337/diacare.24.4.643. PMID 11315823
- [Background] Diabetes Research in Children Network (DirecNet) Study Group; Tsalikian E, Kollman C, Tamborlane WB, Beck RW, Fiallo-Scharer R, Fox L, Janz KF, Ruedy KJ, Wilson D, Xing D, Weinzimer SA. Prevention of hypoglycemia during exercise in children with type 1 diabetes by suspending basal insulin. Diabetes Care. 2006 Oct;29(10):2200-4. doi: 10.2337/dc06-0495. PMID 17003293
- [Derived] Rickels MR, DuBose SN, Toschi E, Beck RW, Verdejo AS, Wolpert H, Cummins MJ, Newswanger B, Riddell MC; T1D Exchange Mini-Dose Glucagon Exercise Study Group. Mini-Dose Glucagon as a Novel Approach to Prevent Exercise-Induced Hypoglycemia in Type 1 Diabetes. Diabetes Care. 2018 Sep;41(9):1909-1916. doi: 10.2337/dc18-0051. Epub 2018 May 18. PMID 29776987

RESULTS

PARTICIPANT FLOW:
Groups:
- MIni-dose Glucagon Crossover Trial: Each participant will undergo four aerobic exercise sessions (in random order) of a) a Control Trial: Fasted exercise, no basal insulin reduction; b) Strategy 1: Fasted exercise, basal insulin reduction only (50% reduction in basal rate five minutes before exercise, for the duration of the exercise); c) Strategy 2: Fasted exercise, no basal adjustment + pre-exercise and mid-exercise glucose tabs (buccal route-40 grams in total); d) Strategy 3: Fasted exercise, no basal adjustment + pre-exercise mini-dose glucagon (sc). Each period includes 0-165 minutes in the lab and the participant continues to wear a continuous glucose monitor during the afternoon, overnight, and through noon the following day.
Period: Control
Arm/Group | MIni-dose Glucagon Crossover Trial
Started | 16
Completed | 16
Not Completed | 0
Period: Basal Insulin Reduction
Arm/Group | MIni-dose Glucagon Crossover Trial
Started | 16
Completed | 16
Not Completed | 0
Period: Glucose Tabs
Arm/Group | MIni-dose Glucagon Crossover Trial
Started | 16 (16 participants were randomized but only 15 completed all 4 periods.)
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Glucagon Injection
Arm/Group | MIni-dose Glucagon Crossover Trial
Started | 16 (16 participants were randomized but only 15 completed all 4 periods.)
Completed | 15
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all patients who completed the crossover trial.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [25 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Type 1 Diabetes Duration, Continuous [Median (Inter-Quartile Range); unit: years] | 22 [14 to 31]
HbA1c [Median (Inter-Quartile Range); unit: %] | 6.8 [6.5 to 7.6]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 24 [23 to 27]
VO2Max [Median (Inter-Quartile Range); unit: mL/kg/min] | 42 [35 to 51]

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Response During Exercise and Early Recovery
Description: Comparison of glycemic response (from blood glucose) during exercise and early recovery between each exercise strategy.
Time Frame: 0 to 75 minutes following exercise initiation (0, 5, 10, 15, 25, 35, 45, 50, 55, 60, 75 min)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 15 | 15 | 15 | 15
mg/dL
  Plasma Glucose Concentration (End of Exercise) | 86 (30) | 85 (25) | 174 (59) | 161 (39)
  Plasma Glucose Concentration (End Early Recovery) | 90 (34) | 92 (34) | 222 (66) | 163 (49)
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); The mini-dose glucagon (MDG) condition was compared with each of the conditions. In the event that exercise was terminated early due to glucose <70 mg/dL and the participant was treated for hypoglycemia (or if participant was treated for hypoglycemia during early recovery [prior to the meal]), the nadir glucose value was carried forward through the end of early recovery; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mixed model w/ repeated measures to account for correlation from cross-over design and multiple measures, adjusting for baseline glucose and period

2. Secondary Outcome: Number of Participants With Hypoglycemia (<70 mg/dL) During Exercise and Early Recovery
Description: Comparison of occurrence of hypoglycemia (<70 mg/dL from blood glucose) during exercise and early recovery between each exercise strategy.
Time Frame: 0 to 75 minutes following exercise initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 6 | 5 | 0 | 0
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Other; p = 0.99, Mixed Models Analysis; Adjusted for subject effect, exercise session, and baseline blood glucose

3. Secondary Outcome: Number of Participants With Hyperglycemia (≥250 mg/dL) During Exercise and Early Recovery
Description: Comparison of occurrence of hyperglycemia (≥250 mg/dL from blood glucose) during exercise and early recovery between each exercise strategy.
Time Frame: 0 to 75 minutes following exercise initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 5 | 1
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.15, Mixed Models Analysis; Adjusted for subject effect, exercise session, and baseline blood glucose

4. Secondary Outcome: Continuous Glucose Monitor (CGM) Metrics During Late Recovery - Nadir Glucose
Description: Comparison of nadir glucose from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
mg/dL | 45 [39 to 60] | 44 [40 to 56] | 49 [40 to 55] | 51 [40 to 53]
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.99, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

5. Secondary Outcome: CGM Metrics During Late Recovery - Peak Glucose
Description: Comparison of peak glucose from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
mg/dL | 241 [216 to 279] | 239 [222 to 299] | 267 [211 to 331] | 269 [235 to 281]
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.43, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

6. Secondary Outcome: CGM Metrics During Late Recovery - Mean Glucose
Description: Comparison of mean glucose from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
mg/dL | 129 [114 to 144] | 139 [127 to 149] | 130 [117 to 148] | 147 [126 to 161]
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.16, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

7. Secondary Outcome: CGM Metrics During Late Recovery - Coefficient of Variation
Description: Comparison of the coefficient of variation from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
percentage | 32 [29 to 42] | 35 [33 to 40] | 36 [32 to 42] | 33 [31 to 35]
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.69, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

8. Secondary Outcome: CGM Metrics During Late Recovery - Time < 54 mg/dL
Description: Comparison of percentage of time < 54 mg/dL from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
percentage | 3 (3) | 3 (3) | 3 (1) | 2 (2)
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.67, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

9. Secondary Outcome: CGM Metrics During Late Recovery - Time < 70 mg/dL
Description: Comparison of percentage of time < 70 mg/dL from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
percentage | 10 (9) | 8 (6) | 8 (6) | 6 (4)
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.84, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

10. Secondary Outcome: CGM Metrics During Late Recovery - Time in Range (70-180 mg/dL)
Description: Comparison of percentage of time in range (70-180 mg/dL) from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
percentage | 73 (12) | 71 (10) | 69 (20) | 67 (15)
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.63, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

11. Secondary Outcome: CGM Metrics During Late Recovery - Time > 180 mg/dL
Description: Comparison of percentage of time > 180 mg/dL from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
percentage | 16 (13) | 21 (12) | 23 (20) | 26 (16)
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.24, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

12. Secondary Outcome: CGM Metrics During Late Recovery - Time > 250 mg/dL
Description: Comparison of percentage of time > 250 mg/dL from CGM between the exercise strategies.
Time Frame: 90 min after the standard meal until 1200 noon the day after each exercise session
Population: Included data were limited to periods with at least 12 hours of CGM data
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
Number analyzed (Participants) | 14 | 13 | 13 | 14
percentage | 1 (2) | 4 (9) | 9 (17) | 5 (7)
Statistical Analysis 1: Comparison: Control vs Basal Insulin Reduction vs Glucose Tabs vs G-Pen Mini™ (Glucagon Injection); Test type: Superiority; p = 0.26, Mixed Models Analysis; Accounted for correlation due to cross-over design and adjusted for exercise session

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) were collected 12 hours prior to each exercise session, during each exercise session, and during the day after each exercise session.
Description: Hypoglycemia, hyperglycemia, injection-related, and exercise-induced events only reported as AEs when criteria below met.
  Hypoglycemia: event required dextrose or glucagon to treat; Hyperglycemia: evaluation or treatment obtained from a health care provider or event involved Diabetic Ketoacidosis; Injection-related events: treatment was given; Exercise-induced events: subject falls or has signs of heart attack, poor perfusion, angina, pathologic arrhythmia, or other condition not expected
Arm/Group | Control | Basal Insulin Reduction | Glucose Tabs | G-Pen Mini™ (Glucagon Injection)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02660242/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT02660242/SAP_001.pdf